CLINICAL TRIAL: NCT06202599
Title: Fruquintinib-based Treatment for Refractory Bone and Soft Tissue Sarcomas After Several Lines of TKIs' Resistance:A Multicenter Retrospective Study
Brief Title: Fruquintinib-based Treatment for Refractory Bone and Soft Tissue Sarcomas After Several Lines of TKIs' Resistance
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Principal Investigator, Peking University People's Hospital
Other Study IDs: PKUPH-sarcoma 17
Record Dates: First submitted 2023-12-21; First posted 2024-01-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Bone Sarcoma; Soft Tissue Sarcoma; Refractory Tumor
Keywords: Fruquintinib; Osteosarcoma; Ewing sarcoma; Soft Tissue Sarcomas; TKIs
MeSH Terms: conditions — Bone Neoplasms; Sarcoma; Neoplasms; Osteosarcoma; Sarcoma, Ewing | interventions — HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Fruquintinib treatment group
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — For patients with pulmonary metastasis only, we mostly gave them fruquintinib with 7 mg in adults and 3-5 mg in children (<10 years) orally per day (5 days on and 2 days off). If patients were extrapulmonary metastasis, we usually used combinations with metronomic chemotherapy (2/3 or 3/5 or even 1/2 of the usual dose) or immunotherapy.

SUMMARY:
This multicenter retrospective study assessed the efficacy and safety of fruquintinib-based treatment in patients with refractory bone and soft tissue sarcomas after several lines of TKIs' resistance.

DETAILED DESCRIPTION:
The short-lived duration of disease control and secondary drug resistance have posed a threat to the effect of TKIs. Fruquintinib is a novel TKI with a high selectivity of VEGFR-1,2,3 without metabolism by liver enzymes and was approved for application in mCRC. Serious drug resistance and the unique characteristics of fruquintinib have prompted us to verify whether this drug can reverse TKIs' resistance at a higher dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed bone or soft tissue sarcomas;
2. Progressed after several lines of therapy;
3. Previously treated with other TKIs before fruquintinib;
4. Received fruquintinib-based treatment;
5. Measurable lesions according to the Response Evaluation Criteria for Solid Tumors (RECIST) version1.1;
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤3

Exclusion Criteria:

1. Failure to complete regular follow-up after administration.
2. Discontinued the fruquintinib-based treatment due to neither progression nor unacceptable toxicity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received fruquintinib-based treatment with refractory bone and soft tissue sarcomas in Peking University People's Hospital and The Second Affiliated Hospital ZheJiang University School of Medicine was included.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
PFS | 4months
  The time from the first administration of fruquintinib to the date of first documentation of disease progression or death, whichever occurred first.

SECONDARY OUTCOMES:
OS | 1year
  OS was calculated from the use of fruquintinib until death from any cause
ORR | 1year
  ORR was defined as the proportion of patients with the best overall response of complete or partial response(CR+PR) according to the Response Evaluation Criteria for Solid Tumors(RECIST) version 1.1.
DCR | 1year
  DCR was defined as the proportion of patients with the best overall response of complete or partial response or stable disease(CR+PR+SD) according to RECIST 1.1.
AEs | 1year
  AEs were graded and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events(CTCAE ) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Xie, M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No